CLINICAL TRIAL: NCT05903469
Title: Implicit and Explicit Assessment of Suicide Risk
Acronym: MIERIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier Pinel d'Amiens (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0118
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Implicit Association Test; Suicide; Prevention, Suicide; Suicide Risk Factor
Keywords: Implicit association test; Suicide; Prevention, Suicide; suicide risk factor
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patient with explicit suicidal ideation and suicide attempt (Experimental)
  Interventions: Other: Implicit Attitude Test
- Patient with explicit suicidal ideation without suicide attempt (Experimental)
  Interventions: Other: Implicit Attitude Test
- Patient without explicit suicidal ideation (Active Comparator)
  Interventions: Other: Implicit Attitude Test

INTERVENTIONS:
Other: Implicit Attitude Test — The IAT (Implicit Attitude Test) is a method of indirectly measuring the relative strength of associations between different concepts stored in memory based on reaction times on computer. The general idea behind this measure is that an individual will be much faster to categorize an object into a predetermined category, if this categorization is consistent with their own way of processing information.

SUMMARY:
In 2007 Nock & Banaji developed a so-called implicit suicide risk measurement using a computer tool: the Implicit Association Test (IAT). This measurement, associated with traditional evaluations, makes it possible to better predict suicidal recurrence. In 2020, the Poitiers team of Tello was able to replicate these results on a French population. However, although a high IAT score predicts the onset of suicide at 1 year, there is no data on how this score changes over time nor even data concerning the measure's ability to differentiate a population with explicit suicidal ideation from a population without explicit suicidal ideation. The investigators therefore seek to demonstrate an evolution of implicit suicidal ideation over time by replicating the measurement at inclusion, at 6 months and at 12 months, for different patient profiles: Suicidal ideation vs No suicidal ideation and suicide attempt vs no suicide attempt. Patients will be recruited from the emergency-unit of CHU Amiens-Picardie and will take the suicide-IAT as well as various questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Person presenting to emergencies for psychiatric reasons
* Adult person
* Free and informed consent signed
* Person speaking and writing French fluently

Exclusion Criteria:

* Neurological disorders or major cognitive deterioration: presence of confusion
* Acute psychotic decompensation
* Troubled acute behavior
* Abuse Impregnation of a toxic substance and / or drug impairing cognitive functions at the time of assessment
* Adult under protective measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Variation of IAT score betwenn the 3 groups | one year
  IAT is Implicit Attitude Test The IAT is a brief computer-administered test that uses people's reaction times when classifying semantic stimuli to measure the automatic mental associations they hold about various topics, in this case, life and death/suicide. The death/suicide IAT will be administered and scored in keeping with standard IAT procedures. Response latencies for all trials were recorded and analyzed using the standard IAT scoring algorithm.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No